CLINICAL TRIAL: NCT01587430
Title: Multicenter Randomised Clinical Trial in Acute Myeloid Leukemia Treatment Based on Three Anthracyclines, Comparing Two Types of Consolidation With Different ARA-C Doses Followed by One Year Maintenance
Brief Title: 3 Anthracyclines, 2 Types of Consolidation With Different ARA-C Doses and Maintenance in Adult Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, MD PhD, National Research Center for Hematology, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML-01.10
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; anthracyclines; high dose cytarabine; maintenance
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose ARA-C (Active Comparator): High dose ARA-C will be applied after two 7+3 induction courses during the first and the second consolidation courses: ARA-C 1 g/m2 bid 1-3 days with idarubicin (8mg/m2 3-5 days)and mitoxantrone (10 mg/m2 3-5 days)
  Interventions: Drug: high dose ARA-C
- standard dose ARA-C (Active Comparator): Standard dose ARA-C will be applied after two 7+3 induction courses the first and the second consolidation courses : ARA-C 100 g/m2 bid 1-7 days with idarubicin (8mg/m2 1-3 days)and mitoxantrone (10 mg/m2 1-3 days)
  Interventions: Drug: standard dose ARA-C

INTERVENTIONS:
Drug: high dose ARA-C — high dose ARA-C consolidation together with high cumulative dose of anthracyclines daunorubicin, idarubicin, mitoxantrone(720-660 mg/m2)
  Arms: high dose ARA-C
Drug: standard dose ARA-C
  Other Names: standard dose ARA-C consolidation together with high cumulative dose of anthracyclines daunorubicin, idarubicin, mitoxantrone(720-660 mg/m2)
  Arms: standard dose ARA-C

SUMMARY:
The goal: to evaluate the role of high dose ara-c plus idarubicin and mitoxantrone consolidation followed by maintenance in the setting of high total cumulative anthracyclines dose(720-660 mg/m2).

DETAILED DESCRIPTION:
In previous Russian AML multicenter studies it was shown that escalation of ARA-C dose (from 5,6 g to 72 g in 4 induction/consolidation courses) in parallel with anthracyclines dose reduction (from 630 mg/m2 to 285 mg/m2)did not improve survival, but decreased feasibility. In the ongoing trial we try to learn whether anthracyclines dose escalation (up to 720-660 mg m2) will or will not equivalise the standard (5,6 g in 4 induction/consolidation courses) and high (14,8 g) ARA-C doses.

ELIGIBILITY:
Inclusion Criteria:

* de novo acute myeloid leukemia - age 15-60

Exclusion Criteria:

* secondary acute myeloid leukemia
* acute myeloid leukemia from myelodysplastic syndrome
* Ph+ acute myeloid leukemia

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 245 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-04 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Valeriy G Savchenko, Study Director — National Research center of Hematology
Locations (1):
- National Research Center for Hematology, Moscow, Russia

REFERENCES:
- [Derived] Parovichnikova EN, Troitskaia VV, Kliasova GA, Kuz'mina LA, Sokolov AN, Paramonova EV, Galstian GM, Kessel'man SA, Drokov MIu, Vasil'eva VA, Obukhova TN, Kulikov SM, Savchenko VG. [Treating patients with acute myeloid leukemias (AML) according to the protocol of the AML-01.10 Russian multicenter randomized trial: the coordinating center's results]. Ter Arkh. 2014;86(7):14-23. Russian. PMID 25314773